CLINICAL TRIAL: NCT00512421
Title: Phase 2 Study of Computer Assisted Surgery vs Conservative Surgery- Accuracy Study.
Brief Title: Navigated EM Total Knee Replacement: Accuracy Study
Status: Terminated | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: LIB002-HMO-CTIL
Record Dates: First submitted 2007-08-05; First posted 2007-08-07 (Estimated); Last update posted 2011-09-16 (Estimated); Status verified 2011-08

CONDITIONS: Total Knee Replacement
MeSH Terms: interventions — Surgery, Computer-Assisted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- A: navigation technique
  Interventions: Procedure: computer-assisted surgery
- B: conservative surgery
  Interventions: Procedure: computer-assisted surgery
- C: Historical control

INTERVENTIONS:
Procedure: computer-assisted surgery
  Groups: A; B

SUMMARY:
The use of computer-assisted surgery by orthopedic surgeons experienced in the performance of total knee arthroplasty may result in better overall limb and implant alignment and fewer outliers as compared with the findings after manual total knee arthroplasty.

The alignment results in previous studies were based on radiographic measurements. The sensitivity of radiographic assessment of limb and implant alignment may not be significant enough to distinguish small differences between computer-assisted surgery and manual techniques.

It is possible that alignment differences that were too minor to be exposed on standard radiographs might result in long-term differences in the durability of arthroplasties performed with use of computer-assisted surgery or manual techniques.

Moreover it is possible to measure additional implant positioning parameters with computed tomography (CT) technology.

In this study, the investigators would like to add new method, for accurate measurement of implant alignment and to correlate its results with clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Signing informed consent

Exclusion Criteria:

* Pregnancy
* Soldiers in active military service

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: men and women that are candidates for total knee replacement.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Meir Libergall, Prof., Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Orthopedic Department, Jerusalem, Israel